CLINICAL TRIAL: NCT03594383
Title: Lung Point-of-care Ultrasound for Acute Respiratory Infections in Resource-constrained Settings - a Pilot Study for Training Community Health Workers
Brief Title: Lung Ultrasound for Acute Respiratory Infections by Community Health Workers
Acronym: L-POCUS
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Collaborators: The Hospital for Sick Children (Other); Grand Challenges Canada (Other)
Responsible Party: Principal Investigator, Dr Fatime Mir, Assistant Professor, Aga Khan University
Other Study IDs: 5106-Ped-ERC-17
Record Dates: First submitted 2018-05-03; First posted 2018-07-20 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Child; Pneumonia
Keywords: Lung; POCUS; Pneumonia; ARI; CHWs
MeSH Terms: conditions — Pneumonia | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ULTRASOUND — Lung ultrasound done through POCUS to diagnose pneumonia

SUMMARY:
The specific objectives focus on using a train-the-trainer model to educate CHWs in Pakistan on performing and interpreting pediatric lung POCUS. In the first phase, the POCUS experts from Toronto will rigorously train the first generation of local lung POCUS users who are Pakistani health care providers to become local lung POCUS trainers. These first generation trainers will subsequently collaborate with the POCUS experts from Toronto to develop a two-day training program for lung POCUS image interpretation and acquisition that is tailored to novice users (CHWs) in low-resource settings. In the second phase, the first generation local lung POCUS trainers will deliver and evaluate the new training program to the second generation of users - a group of CHWs in Karachi. In the third phase, we will establish the reliability of CHWs to perform lung POCUS on pediatric patients with respiratory symptoms, upon completion of the training program developed by local trainers.

DETAILED DESCRIPTION:
POCUS is an example of technologies that are moving out of hospitals and to the point-of-care. The true potential of these novel diagnostics to improve global pediatric pneumonia outcomes will only be realized if they can be employed by CHWs in community settings in LMICs. No work has yet focused on the performance of POCUS by non-medically-trained CHWs in LMICs. Demonstrating that accurate POCUS performance and interpretation can be achieved by non-medically-trained CHWs after focused and succinct training is the first step towards developing a novel pediatric pneumonia diagnosis and management algorithm for LMICs. Feedback from these ultrasound-naïve users about their lung POCUS learning experience is also needed to clarify which POCUS findings would be best suited to this algorithm.

The research team in AKUH will recruit and consent interested CHWs from AKU field sites in Karachi. The target is to recruit a convenience sample of 3 CHWs, who will be as representative as possible of the experience and skill sets as the average CHW in a government program. Study participants will be identified and approached by clinical team members in the AKUH emergency department, outpatient clinic and pediatric ward.

Triaging children with ARI into accurate treatment categories will lead to increased paediatric pneumonia survival, improved antibiotic stewardship, and more appropriate resource use, all of which are clinically and programmatically significant in highest disease burden settings. This project also lays the foundation for future projects that harness the trans-formative potential of POCUS for global child health.

ELIGIBILITY:
Children between the ages of 2 to 59 months who is presenting with at least one of the following in the last 72 hours:

* patient reported symptoms (cough, coryza, reported fast breathing) AND
* WHO CRITERIA (FAST BREATHING (≥50 /min age if 2-12months, ≥40/min if age 1-5years) AND/OR CHEST INDRAWING and DANGER SIGNS (unable to drink, persistent vomiting, convulsions, lethargic or unconscious, stridor in a calm child, severe malnutrition) AND/ OR STRIDOR
* AND/OR Oxygen saturation < 96% OR CXR/CT pneumonia OR MD diagnosed pneumonia ● Patients admitted for non-respiratory symptoms may be included in the absence of exclusion criteria (this group will only be considered for the study if interim analysis reveals low recruitment of patients with a normal lung POCUS appearance)

Exclusion criteria:

* patients that previously underwent lung POCUS by the same lung POCUS operator during the same visit to AKUH
* chest tube insertion or video-assisted thoracoscopic surgery (VATS) during the current visit to AKUH (since the equipment in situ and/or dressing might bias POCUS interpretation)
* inability to understand informed consent

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between age of 2 months to 5 years and presenting with signs and symptoms of pneumonia, will be identified and approached by clinical team members in the AKUH emergency department, outpatient clinic and pediatric ward. The research member will review the study with the family and obtain informed consent from parents.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
primary outcome of interest will be the inter-rater reliability of lung POCUS findings (on a cohort of patients at AKUH with ARI) between the newly trained CHWs and a local lung POCUS trainer. | 12 months
  Proportion of CHWs undergoing training in lung POCUS with a passing score 80% in a computer-based test (consisting of 60 lung POCUS video clips) with questions to determine their image interpretation skills as a reflection of technical performance. On completion of training program, they will perform lung POCUS on pediatric patients presenting to Aga Khan University Hospital (AKUH) with respiratory symptoms.
  For primary outcome of inter-rater reliability, the Cohen's kappa statistic will be calculated using standardized formulas. in the end will be describing the kappa statistic between final interpretations (overall and for each lung zone) of each scan by the CHWs as compared to the POCUS expert.

SECONDARY OUTCOMES:
Train the trainer | 20 days
  the assessment of the first generation local lung trainers will include:
  1. a computer-based test with 60 questions as an indication of general knowledge pertaining to lung POCUS
  2. OSATS as indication of their technical performance
  3. 5 mentored scans observed by POCUS experts
  4. 20 lung scans with quality assurance performed by POCUS experts
  Upon completion of the Train the trainer phase, the first generation users will be deemed qualified local lung POCUS trainers. Subsequently, these new trainers will collaborate with the POCUS experts from Toronto to develop training program B, which will be modified to target novice non-physician users.
Train novice users | 2 days
  1. Performance assessment of the CHWs upon completion of training program B delivered by local lung POCUS trainers:
     1. CHWs' scores on a newly developed computer-based test (consisting of 60 lung POCUS video clips) as an indication of their image interpretation skills
     2. CHWs' scores on a checklist titled Observed Structured Assessment of Technical Skills (OSATS) as a reflection of technical performance in POCUS
  2. Program evaluation (descriptive feedback) of training program B provided by CHWs
  Proportion of CHWs undergoing training in lung POCUS with a passing score 80% in a computer-based test (consisting of 60 lung POCUS video clips) with questions to determine their image interpretation skills as a reflection of technical performance. On completion of training program, they will perform lung POCUS on pediatric patients presenting to Aga Khan University Hospital (AKUH) with respiratory symptoms.
Reliability of CHW lung POCUS use on children with acute respiratory illnesses | 6 months
  1. Raw agreement between:
     1. POCUS findings of CHWs and chest x-ray findings (if performed)
     2. POCUS findings of CHWs and final diagnosis in chart
     3. Chest x-ray findings (if performed) and final diagnosis in chart
  2. Descriptive feedback of the CHWs' user experience of lung POCUS
  POCUS recordings (with no patient identifiers) will be made for each patient scan performed by the CHWs. These clips will be captured via the Lumify device and uploaded to a computer and then to an online server, from which a blinded pediatric lung POCUS expert in Toronto can download and perform the quality assurance check. This second expert will not have participated in the study intervention phase at AKUH.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Mir, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan